CLINICAL TRIAL: NCT03361241
Title: Comparison of Effects of Training in a Virtual Environment With and Without Physiotherapeutic Intervention on the Motor Function, Postural Control and Gait in Chronic Stroke Patients : A Randomized Controlled Trial
Brief Title: Comparison of Training in Virtual Environment With and Without Physiotherapeutic Intervention in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USPCR001
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: Stroke; Postural Balance; Motor Function; Gait; Virtual Reality Exposure Therapy; Physiotherapist
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single blinded (outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Physiotherapeutic Intervention (Experimental): Virtual reality training without physiotherapeutic intervention
  Interventions: Other: No Physiotherapeutic Intervention
- Physiotherapeutic Intervention (Active Comparator): Virtual reality training with physiotherapeutic intervention
  Interventions: Other: Physiotherapeutic Intervention

INTERVENTIONS:
Other: No Physiotherapeutic Intervention — Experimental group will perform a balance training program in a virtual environment (using a gaming system with balance board device - eight games of Nintendo Wii Fit®, for 14 sessions) without verbal/manual physiotherapeutic intervention.
  Initially, instructions about the rules and strategies of how to play the game and control the avatar will be provided.
  Then the patient will be invited to start the game, and in the two attempts of the training no manual or verbal assistance will be provided. Physiotherapist participation during training will be restricted to ensuring patient safety, providing motivational verbal stimuli, and replicating the feedback provided by the game at the end of each attempt.
  Other Names: Experimental Group
  Arms: No Physiotherapeutic Intervention
Other: Physiotherapeutic Intervention — Control group will perform a balance training program in a virtual environment (gaming system with balance board device - eight games of Nintendo Wii Fit®, for 14 sessions) with verbal and manual physiotherapeutic intervention. Initially, instructions about the rules and strategies of how to play the game and control the avatar will be provided. Then the patient will be invited to start the game, and in the first attempt of the training physiotherapist will provide manual and verbal assistance, providing corrections on movement (avoiding compensatory movements). In the second attempt, no manual or verbal assistance will be provided (only ensuring patient safety, providing motivational verbal stimuli), allowing the patient to organize his or her performance.
  Other Names: Control Group
  Arms: Physiotherapeutic Intervention

SUMMARY:
The aim of this study is to compare the effects of balance training in a virtual environment with and without physiotherapeutic intervention on the motor function, balance and gait in chronic stroke patients.

It is a prospective, single blinded, randomized clinical trial performed at Center of Research of the Department of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University. Forty patients will be randomly assigned in control and experimental group.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of a balance training program in a virtual environment (using a gaming system with balance board device) with and without verbal/manual physiotherapeutic intervention, on the motor function, balance and gait in chronic stroke patients.

It is a prospective, single blinded, randomized clinical trial, performed at Center of Research of the Department of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University.

Forty chronic stroke patients will be randomly in control and experimental group, 20 each one. Both groups conduct 14 training sessions, twice a week, for seven weeks. Each session will consist a 30 minute-global-exercise series including stretching, muscle strength and axial mobility exercises. After this, both groups will perform more 30 minutes of balance training using eight Wii Fit games which stimulate motor and cognitive functions.

The main outcome measures will be: the lower limb subscale of the Fugl-Meyer Assessment (FMA-LE); Balance Evaluation Systems Test (BESTest) and 6- minute walk test (6MWT).

ELIGIBILITY:
Inclusion Criteria:

* hemiparetic status resulting from a single stroke at least 6 months earlier;
* the ability to walk 10 m independently with or without an assistive device;
* a Montreal Cognitive Assessment (MoCA) score of ≥ 20;
* the absence of a musculoskeletal condition that could potentially affect the ability to stand or walk safely;
* the absence of serious visual impairment or a hearing disorder;
* muscle strength ≥ 3 in lower limbs;
* ability to understand and follow simple instructions.

Exclusion Criteria:

* severe dementia or aphasia;
* hemispatial neglect, ataxia or any other cerebellar symptom;
* inability to stand without minimal assist;
* uncontrollable medical complications
* participation in other studies or rehabilitation programs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Balance Evaluation Systems Test (BESTest) | Up to 3 months
  Balance Evaluation Systems Test (BESTest) measures balance. It includes 36 items that evaluate performance of 6 balance systems: biomechanical constraints, stability limits/verticality, anticipatory postural adjustments, postural responses, sensory orientation, and stability in gait.

SECONDARY OUTCOMES:
The lower limb subscale of the Fugl-Meyer Assessment (FMA-LE) | Up to 3 months
  FMA-LE is a subscale measuring lower limb motor recovery. It examines movement and coordination of the hip, knee, and ankle in the supine, sitting, and standing positions. Each item is scored on a 3-point scale (0, cannot perform; 1, partially performs; 2, performs fully). The score range is 0 to 34, with higher scores indicating better lower limb motor performance
6-minute walk test | Up to three months
  The 6MWT is a practical simple test. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). The 6MWT has been used as a measure of functional status of patients.
Limits of Stability | Up to 3 months
  The Limits of Stability subtest quantifies the maximum distance a person can intentionally displace their center of pressure (COP) from start position of midline COP centered over the base of support to eight targets. Location and movement of the COP was indicated by a cursor display projected on a screen in front of the subject. As targets were highlighted, the subject was to move the COP cursor quickly and accurately as possible towards a target located on the Limits of Stability perimeter and hold position as close to the target as possible. The parameters include COP movement velocity and directional control (% to target).
Rhythmic Weight Shift | Up to three months
  The Rhythmic Weight Shift quantifies the subject's active weight shift ability by moving the COP cursor to match velocity and direction of a moving visual target in the medial- lateral (ML) and anterior-posterior (AP) directions at three different velocities.
Stroke Speciﬁc quality of life scale | Up to three months
  Stroke Quality of Life Scale is a self-report assessment that includes 12 stroke subscales with 49 items. The Stroke Speciﬁc Quality of Life Scale attempts to capture the domains of stroke QOL that are insufficiently assessed with generic QOL measures. The 12 subscales, which are unidimensional, are Energy, Family Role, Language, Mobility, Mood, Personality, Self-Care, Social Roles, Thinking, Upper Extremity Function, Vision, and Work-Productivity. Participants responded to each item on a 5-point scale. Domain scores are the averages of the item scores, and the total score is the average of the domain scores. All summary scores therefore range from 1 to 5. Higher scores indicate better function.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PT, PhD, Study Director — University of Sao Paulo; Mariana A Lourenço, PT,Ms Student, Principal Investigator — University of Sao Paulo; Tatiana P Oliveira, PT,PhD Student, Principal Investigator — University of Sao Paulo; Camila S Miranda, PT, MS, Principal Investigator — University of Sao Paulo
Locations (1):
- Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy, School of Medicine, University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamson J, Beswick A, Ebrahim S. Is stroke the most common cause of disability? J Stroke Cerebrovasc Dis. 2004 Jul-Aug;13(4):171-7. doi: 10.1016/j.jstrokecerebrovasdis.2004.06.003. PMID 17903971
- [Background] Borghese NA, Pirovano M, Lanzi PL, Wuest S, de Bruin ED. Computational Intelligence and Game Design for Effective At-Home Stroke Rehabilitation. Games Health J. 2013 Apr;2(2):81-88. doi: 10.1089/g4h.2012.0073. PMID 24761321
- [Background] Broeren J, Claesson L, Goude D, Rydmark M, Sunnerhagen KS. Virtual rehabilitation in an activity centre for community-dwelling persons with stroke. The possibilities of 3-dimensional computer games. Cerebrovasc Dis. 2008;26(3):289-96. doi: 10.1159/000149576. Epub 2008 Jul 31. PMID 18667809
- [Background] Laver K, George S, Thomas S, Deutsch JE, Crotty M. Cochrane review: virtual reality for stroke rehabilitation. Eur J Phys Rehabil Med. 2012 Sep;48(3):523-30. Epub 2012 Jun 20. PMID 22713539
- [Background] Laufer Y, Dar G, Kodesh E. Does a Wii-based exercise program enhance balance control of independently functioning older adults? A systematic review. Clin Interv Aging. 2014 Oct 23;9:1803-13. doi: 10.2147/CIA.S69673. eCollection 2014. PMID 25364238
- [Background] Mancini M, Horak FB. The relevance of clinical balance assessment tools to differentiate balance deficits. Eur J Phys Rehabil Med. 2010 Jun;46(2):239-48. PMID 20485226
- [Background] Yatar GI, Yildirim SA. Wii Fit balance training or progressive balance training in patients with chronic stroke: a randomised controlled trial. J Phys Ther Sci. 2015 Apr;27(4):1145-51. doi: 10.1589/jpts.27.1145. Epub 2015 Apr 30. PMID 25995576
- [Background] Dong Y, Sharma VK, Chan BP, Venketasubramanian N, Teoh HL, Seet RC, Tanicala S, Chan YH, Chen C. The Montreal Cognitive Assessment (MoCA) is superior to the Mini-Mental State Examination (MMSE) for the detection of vascular cognitive impairment after acute stroke. J Neurol Sci. 2010 Dec 15;299(1-2):15-8. doi: 10.1016/j.jns.2010.08.051. PMID 20889166
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Horak FB, Wrisley DM, Frank J. The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther. 2009 May;89(5):484-98. doi: 10.2522/ptj.20080071. Epub 2009 Mar 27. PMID 19329772
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Williams LS, Weinberger M, Harris LE, Clark DO, Biller J. Development of a stroke-specific quality of life scale. Stroke. 1999 Jul;30(7):1362-9. doi: 10.1161/01.str.30.7.1362. PMID 10390308

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03361241/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03361241/ICF_001.pdf